CLINICAL TRIAL: NCT07317024
Title: Additional Effects of Shockwave Therapy Along With Median Nerve Gliding Exercises in Patient With Carpal Tunnel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/11
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS); Mobility; Hand Functions
Keywords: Carpel Tunnel Syndrome; Shockwave Therapy; Nerve Gliding Exercises; NCS; Nerve Velocity; Nerve Amplitude; Pain; Functional strength
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTIONAL GROUP B- SHOCKWAVE THERAPY WITH NERVE GLIDING (Experimental): The participants will recieve 3 minutes of Shockwave therapy along with nerve gliding exercises thrice a week for 4 weeks with total 30 minutes sessions.
  Intensity of exercise will be incresed gradually and according to patient progress with break time to avoid fatigue.
  The intensity of the shock waves is set at 0.03 mJ/mm².The applied pressure is around 1.6 bar. Each session involves deliver in 2000 shocks. Shockwave therapy will targeted at the area between the thenar and hypothenar eminences on the palm
  Interventions: Procedure: SHOCKWAVE THERAPY
- CONTROL GROUP A- CONVENTIONAL PHYSICAL THERAPY (Active Comparator): The participants will perform nerve gliding exercises in which hand and wrist will moved through six more positions to mobilize the median nerve. Subjects will recieve protocal of 30 mins thrice a week for 4 weeks with 2 min rest in between.
  The exercises will focus on mobility of median nerve and reduce compression related symptoms to improve function and strength.
  Interventions: Procedure: NERVE GLIDING EXERCISES

INTERVENTIONS:
Procedure: NERVE GLIDING EXERCISES — Median nerve mobilization involves exercises aimed at relieving pressure in the carpal tunnel, making it a common treatment for carpal tunnel syndrome (CTS). Techniques may stretch the nerve from both ends or apply tension to one end while releasing the other. Some techniques stretch the nerve from both ends at the same time, while others apply tension to one end while allowing the other end to relax. Conservative treatment options include Neurodynamic mobilization, which utilizes neural gliding to promote nerve movement in relation to surrounding musculoskeletal tissues. This biomechanical strategy aims to decrease swelling and adhesions within the carpal tunnel, thereby restoring the nerve's mobility. Studies have also reported neuromodulatory effects from neural mobilization techniques due to the chronic nature of CTS.
  Arms: CONTROL GROUP A- CONVENTIONAL PHYSICAL THERAPY
Procedure: SHOCKWAVE THERAPY — Shockwave therapy is a physical intervention intended for diverse musculoskeletal disorders. There are two primary categories: targeted extracorporeal shockwave therapy (ESWT) and radial shockwave therapy. The two approaches vary in their generation, characteristics, and impact. Extracorporeal Shock Wave Therapy (ESWT) is generated in water via electrohydraulic, electromagnetic, or piezoelectric sources. This technique generates a concentrated pressure field that converges at a profound focal point, yielding maximum pressure. Conversely, radial shockwaves are produced by propelling a projectile through an air-compressed tube, resulting in a diverging pressure field that affects the tissue more superficially. ESWT in carpal tunnel syndrome (CTS) have reported enhancements in symptoms, functional scores and pain levels. Additionally, low-to-moderate intensity ESWT has been shown to have positive effects on nerve conduction studies.
  Arms: INTERVENTIONAL GROUP B- SHOCKWAVE THERAPY WITH NERVE GLIDING

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a widespread condition resulting from the compression of the median nerve, causing significant pain, numbness, and weakness in the hand.This study decisively evaluates the impactful effects of integrating shockwave therapy (ESWT) with median nerve gliding exercises.The primary goals are to enhance median nerve function, improve hand performance, and achieve superior pain management.This will be a rigorous non-blinded randomized control trial involving two groups formed through purposive sampling .A total of 12 sessions of shockwave therapy with median nerve gliding exercises and 12 sessions of median nerve gliding exercises were performed in both groups, with three sessions each week over a four-week period. The experimental group were received shockwave therapy and median nerve gliding exercises while the control group were given physical therapy and median nerve gliding exercises.Outcomes will be measured using NCS BTCQ and NPRS. The study will take place over one year at FFH and FUCP, with ethical approval from ERC FUMC.

DETAILED DESCRIPTION:
OBJECTIVE:

The objectives of this study are:

1. To evaluate and compare the effects of shockwave therapy combined with nerve gliding exercises against nerve gliding exercises alone on the velocity and amplitude of the median nerve.
2. To analyze and compare the impact of shockwave therapy combined with nerve gliding exercises versus nerve gliding exercises alone on hand function in individuals with carpal tunnel syndrome.
3. To assess and compare the effects of shockwave therapy combined with nerve gliding exercises with those of nerve gliding exercises alone on reported pain levels.

HYPOTHESIS

Alternate Hypothesis:

There will be statistically significant difference in effects of shockwave therapy combined with nerve gliding exercises and in comparison to nerve gliding exercises alone on hand functional strength, velocity and amplitude of the median nerve and pain. . (p<0.05).

Null Hypothesis:

There will be no statistically significant difference in effects of shockwave therapy combined with nerve gliding exercises and in comparison to nerve gliding exercises alone on hand functional strength, velocity and amplitude of the median nerve and pain. (p<0.05).

Research Design: Experimental study. Randomized Control Trial

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both females and males were included.
* Age: Between 20 and 40 years old.
* Patients exhibiting positive results on the "Phalen's test and Tinel's test."
* Presence of symptoms, including pain, tingling and numbness, affecting the first, second and third fingers.

Exclusion Criteria:

* Individuals with a history of wrist surgery.
* Patients with active infections or cancer, for whom shockwave therapy is contraindicated.
* Pregnant females.
* Individuals diagnosed with rheumatoid arthritis.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Perceived Pain Level | 4 weeks
  The Numeric Pain Rating Scale (NPRS) is a patient-reported measure of pain intensity, with lower scores indicating less pain.
  Scores between 0-1 indicate minimal pain, generally with little to no interference in daily life. Mild pain, characterized by scores of 2-3. A score in the 4-6 range signifies moderate pain, which is noticeable, can interfere with specific daily functions. Finally, severe pain, represented by scores of 7-10, is intense.
Hand Movement and Function | 4 weeks
  Functional Status Scale (BCFSS) measures the difficulty patients experience with performing specific daily activities affected by CTS, also often on a 1-5 point scale, where higher scores reflect greater functional limitation. Lower scores mean better hand function. Scores around 1.0-2.0 indicate mild impact, 2.0-3.0 moderate impact, and above 3.0 severe impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan